CLINICAL TRIAL: NCT00129870
Title: CONCEPT - Phase IV, Randomized, Prospective, Multicenter Comparison of Intermittent Schedule of Oxaliplatin Combined With FOLFOX/Bevacizumab vs Conventional Mode of Administration of FOLFOX/Bevacizumab + Neuroprophylaxis With Calcium/Magnesium for Optimization of First-Line Therapy of Metastatic Colorectal Cancer
Brief Title: CONCEPT: Comparison of Oxaliplatin vs Conventional Methods With Calcium/Magnesium in First-Line Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unplanned interim analysis by DSMB indicated possible reduced response rate with the addition of Ca/Mg in pooled population. Further analysis pending.
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: L_9444
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
The primary rationale for this study is to develop an optimized schedule of administration of FOLFOX + bevacizumab that maximizes the efficacy and safety of this regimen when administered to patients with advanced colorectal cancer. The hypothesis is that the use of an intermittent oxaliplatin (IO) schedule of FOLFOX/bevacizumab will allow these patients to continue on treatment for a longer period of time by reducing the proportion of patients who discontinue therapy early because of treatment-related toxicities and thus increasing the possibility of a longer time to progression.

The primary objective is:

* To test the hypothesis that an intermittent oxaliplatin (IO) schedule of FOLFOX/bevacizumab will allow patients to remain on therapy for a longer period of time compared to a conventional "treat-to-failure" schedule, by reducing the proportion of patients who discontinue therapy for treatment-related toxicities.

The secondary objectives are:

* To evaluate the impact of calcium/magnesium infusions on the incidence and severity of neurotoxicity in subjects receiving either the IO or conventional FOLFOX/bevacizumab treatment schedules as first-line treatment for metastatic colorectal cancer.
* To evaluate the safety and efficacy of the IO versus the conventional schedule + calcium and magnesium infusions, as part of oxaliplatin-based first-line therapy for metastatic colorectal cancer.

ELIGIBILITY:
The following information on clinical trials is provided for information purposes only to allow patients and physicians to have an initial discussion about the trial. This information is not intended to be complete information about the trial, to contain all considerations that may be relevant to potential participation in the trial, or to replace the advice of a personal physician or health professional.

Inclusion Criteria:

* Histologically or cytologically documented metastatic, measurable adenocarcinoma of the colon, rectum, or appendix with no prior therapies for metastatic disease
* ECOG performance status (PS) of 0 or 1
* Adequate hematologic, renal, and hepatic function as defined by required baseline laboratory parameters
* No other serious concomitant disease.

Exclusion Criteria:

* Peripheral neuropathy > Grade 1 at baseline
* History of significant cerebrovascular, cardiovascular, or peripheral vascular disease
* Uncontrolled hypertension (defined as blood pressure > 150/100 mmHg)
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess, within 6 months prior to start of study drug
* Minor surgical procedure, fine needle aspiration, or core biopsy within 7 days prior to start of study drug
* Serious, non-healing wound, ulcer, or bone fracture
* Active gastroduodenal ulcer
* Evidence of bleeding diathesis or coagulopathy
* Significant history of bleeding within 6 months prior to registration
* Prior history of hypertensive crisis or hypertensive encephalopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-02; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure (TTF) for the conventional oxaliplatin (CO) schedule in comparison with the intermittent oxaliplatin (IO) schedule

SECONDARY OUTCOMES:
The incidence of adverse events, including neurotoxicity, as determined using the National Cancer Institute (NCI) Common Toxicity Criteria version 3.0 (CTCAE v3.0)
Quality of life, including oxaliplatin-specific neurologic symptoms determined using the PNQoxali
Tumor response rate (overall and confirmed) based on application of the Response Evaluation Criteria in Solid Tumors (RECIST)
Time to tumor progression (TTP)
Time of tumor control (TTC)
Overall survival (OS)
Reasons for treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Yasir Nagarwala, M.D., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States